CLINICAL TRIAL: NCT01062958
Title: A Retrospective Analysis of Neevo® and Neevo®DHA Compared to a Standard Prenatal Vitamin in Anemia During Pregnancy (N-001)
Brief Title: A Retrospective Analysis of Neevo®/Neevo®DHA Compared to a Standard Prenatal Vitamin in Anemia During Pregnancy
Status: Completed | Type: Observational
Sponsor: Pamlab, Inc. (Industry)
Collaborators: Baylor Health Care System (Other); Women's Clinic Shoals (Unknown); Gainesville Obstetrics & Gynecology (Other); Womens Health Associates (Unknown)
Responsible Party: Sponsor
Other Study IDs: N-001
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Anemia in Pregnancy; Preeclampsia
Keywords: Neevo; Neevo DHA; L-methylfolate; anemia during pregnancy; folic acid; vitamin B12; prenatal vitamins; hemoglobin; iron deficiency; Pregnancy
MeSH Terms: conditions — Pre-Eclampsia; Iron Deficiencies | interventions — Prenatal Care; Folic Acid; Iron; Vitamin B 12

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm #1 (Test group): 50 subjects administered Neevo® or Neevo®DHA daily
  Interventions: Other: Neevo® (a medical food)
- Arm #2 (Control group): 50 subjects administered a prenatal vitamin daily
  Interventions: Other: Prenatal vitamins (≤1mg folic acid, 27 - 35mg iron, and ≤12mcg vitamin B12)

INTERVENTIONS:
Other: Neevo® (a medical food)
  Groups: Arm #1 (Test group)
Other: Prenatal vitamins (≤1mg folic acid, 27 - 35mg iron, and ≤12mcg vitamin B12)
  Groups: Arm #2 (Control group)

SUMMARY:
This study is a multi-site, retrospective chart review to determine the effect of Neevo® or Neevo®DHA (with higher folate and B12) versus standard prenatal vitamins on hemoglobin (Hgb) levels in pregnant women throughout the course of pregnancy. Neevo® is a prescription medical food indicated for the dietary management of women under a doctor's care who face high risk pregnancies, older overactive bladder (OB) patients and patients unable to fully metabolize folic acid. Data will be collected from existing patient charts of subjects administered Neevo® or Neevo®DHA daily compared to subjects administered a prenatal vitamin daily.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females, age 21-39, who received either Neevo®/Neevo®DHA or another standard prenatal vitamin (Prenatal vitamins must contain ≤1 mg folic acid, 27-35mg iron, and ≤12mcg vitamin B12).
* Clinical diagnosis of pregnancy must have been made at ≤12 weeks of pregnancy and on or after January 1, 2008 and delivery must have occurred on or before December 31, 2009.
* Subjects must have been compliant in taking Neevo DHA or other prenatal vitamin.

Exclusion Criteria:

* Subjects should not have taken Prenate®, Prenate®DHA, or Prenate® Elite, which are L-methylfolate-containing prenatal vitamins.
* The following supplements within 2 months prior to randomization; 100mg vitamin C, B12 injection >10mg of B6; >32mg Iron; >1.2mg of folate; an L- methylfolate product that is not a prenatal vitamin such as Life Extension methylfolate, Prothera methylfolate, Thorne 5-MTHF, Metanx®, Neevo®, Neevo®DHA, Deplin®, Cerefolin®, or CerefolinNAC®.
* History of any anemia other than iron deficiency anemia or leukemia.
* Blood transfusion in the 4 months prior to diagnosis of pregnancy.

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Women Who Received Neevo®/Neevo® DHA or Another Standard Prenatal Vitamin
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To determine the effect of Neevo®/Neevo®DHA (with higher folate and B12) versus standard prenatal vitamins on hemoglobin levels in pregnant women throughout the course of pregnancy. | At the time of diagnosis of pregnancy, at Weeks 22-28, and at delivery.

SECONDARY OUTCOMES:
To determine the effect of Neevo®/Neevo®DHA versus standard prenatal vitamins on red blood cell (RBC) levels in pregnant women. | At the time of diagnosis of pregnancy, at Weeks 22-28, and at delivery.
To determine if Neevo®/Neevo®DHA administration during pregnancy results in fewer anemias than with standard prenatal vitamins. | At the time of diagnosis of pregnancy, at Weeks 22-28, and at delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Bentley, CRNP, Principal Investigator — Women's Clinic Shoals
Locations (3):
- United States (3):
  - Women's Clinic Shoals, Sheffield, Alabama
  - Women's Health Associates, Flowood, Mississippi
  - Gainesville Obstetrics & Gynecology, Gainesville, Texas

REFERENCES:
- [Result] Bentley S, Hermes A, Phillips D, Daoud YA, Hanna S. Comparative effectiveness of a prenatal medical food to prenatal vitamins on hemoglobin levels and adverse outcomes: a retrospective analysis. Clin Ther. 2011 Feb;33(2):204-10. doi: 10.1016/j.clinthera.2011.02.010. Epub 2011 Mar 25. PMID 21440300